CLINICAL TRIAL: NCT04112992
Title: An International, Multicenter, Prospective Registry to Investigate Treatment Options and Their Outcomes on Post-traumatic Long Bones Defects
Brief Title: An International, Multicenter, Prospective Registry on Post-traumatic Long Bones Defects
Status: Recruiting | Type: Observational
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: LoBoDe Registry
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Limb Fracture; Bone Loss
Keywords: long bone defect
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Any treatment that is used for a defect of any long bone — Any treatment that is used for a defect of any long bone. All treatments are based on individual clinician's judgement and the patient characteristics. The registry does not dictate any specific treatment.

SUMMARY:
Long bone defect (LBD) is defined as a focalized loss of bone tissue in any long bone of the upper or lower extremity. Long bone defects are a complex problem, that may arise as a complication of many different pathologies, such as trauma, tumors or infection. Whereas post-traumatic defects are the largest group.

Reports estimate that there are almost 4 million bone grafting procedures worldwide per year. However, limb reconstruction in the context of a bony defect is challenging and up to date there is little evidence and treatment recommendations.

In a multi-national approach, the aim of this project is to set up an international, multicenter registry to gather information and details on prevalence or incidence, current treatments, complications and outcome.

DETAILED DESCRIPTION:
The purpose of this project is to set up an international, multicenter registry of patient presenting with defects in long bones. Up to date, treatment remains challenging with little evidenced-based recommendations.

For this purpose, any patient who presents at a study center with a bone defect of the defined expansion of any long bone is eligible for inclusion. Over a 3-year period as many patients as possible are included from the participating sites, at least 600 patients should be included in the registry. Details on any surgical intervention that is used to treat a bone defect will be recorded. Further patient-related and other pre-defined outcome measures will be collected.

There is no formal hypothesis to this registry, hence it will help to identify prevalence and underlying etiologies, evaluate treatment strategies, and highlight possible challenges and complications - and will so help to gather clinical evidence to provide better treatment for patients suffering from a long bone defect.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Skeletally mature
* Post traumatic bone defect > 2 cm either

  * initially after injury or
  * after surgical debridement
* Informed consent obtained, i.e.:

  * Ability to understand the content of the patient information/ICF
  * Willingness and ability to participate in the clinical investigation according to the registry plan
  * Signed and dated EC/IRB approved written informed consent OR
  * Written consent provided according to the IRB/EC defined and approved procedures for patients who are not able to provide independent written informed consent

Exclusion Criteria:

* Any oblique defect that has less than 8cm expansion when adding the defect size of all four cortices
* Any not medically managed severe systemic disease
* Pregnancy
* Prisoners
* Participation in any other medical device or medicinal product registry within the previous 3 months that could influence the results of the present registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a traumatic bone defect in any long bone
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Baseline characteristics | Pre-operative
  Demographics, medical history, comorbidity
Bone defect details | Pre-operative and/or intraoperative
  * Affected bone
  * Localization: Proximal 1/3rd, middle 3rd, distal 1/3rd(for any bone)
  * Size (categorization according Karger classification; definition: a bone defect should be at least 2 cm (Karger Type II)) Type II: 2-5 cm Type III: 5-10 cm Type IV: > 10 cm
Trauma assessment | Pre-operative and/or intraoperative
  * Injury Severity Score (ISS): Grading for each item (points): No injury (0), Minor (1), Moderate (4), Serious (9), Severe (16), Critical (25), Unsurvivable (75)
  * Assessment:
    * Head and neck worst injury
    * Face worst injury
    * Chest worst injury
    * Abdomen worst injury
    * Extremity (including pelvis) worst injury
    * External worst injury
  * Gustilo & Anderson classification for open fractures
    * Type I
    * Type II
    * Type IIIA
    * Type IIIB
    * Type IIIC
  * Tscherne classification for closed fracture and soft-tissue injuries
    * Grade 0
    * Grade 1
    * Grade 2
    * Grade 3
evaluate the bone defect in the context of previous interventions | Intraoperative
  Number of previous interventions: <2, <4, >4
Surgical details & Intraoperative findings 1 | Intraoperative
  * Procedure type:
    * One stage
    * Staged (e.g. Masquelet technique / distraction osteogenesis / bone transport)
    * Ilizarov
  * Bone quality (good, fair, poor) by surgeon's discretion
  * Soft tissue and vascularity (good, fair, poor) by surgeon's discretion
  * Contamination (yes/no)
  Specification:
  * Metal from a bullet
  * Metal from a pole
  * Other Metal
  * Wood
  * Soil
  * Others
    * Surgical time (min)
    * Stabilization technique: Internal device (extra- or intramedullary) / External device (For both, drop down menu will be used)
Surgical details & Intraoperative findings 2 | Intraoperative
  * Bone grafting
    * Autografts
    * Allograft(s)
    * Other synthetics
    * If applicable - time to harvest graft (in minutes)
  * Graft enhancement yes / no
    * Demineralized bone matrix (DBM)
    * Bone morphogenetic protein (BMP)
    * Stem cells
    * Platelet rich plasma (PRP)
    * Other
  * Soft-tissue / vascular / microsurgical procedure yes / no
    * Skin graft
    * Local flap
    * Free flap
  * Additional treatment
    * Systemic antibiotic treatment yes / no
    * Local antibiotic treatment yes / no
    * Post-operative use of a negative pressure dressings (NPWT) or vacuum-assisted closure (VAC) system yes / no
Functional Outcome | 6 months follow-up / 12 months follow-up and/or 6 months after bone union (max 12 months)
  - Assessment of limb function and loss of length
  * Definition: anatomic shortening of the limb in comparison to the contralateral side
  * Assessment in cm
  * Any orthotic used to equalize leg length
Patient related outcome / Quality of life 1 | Screening / 6 months follow-up / 12 months follow-up and/or 6 months after bone union (max 18 months)
  Patient-Reported Outcomes Measurement Information System (PROMIS)
  * Physical function: This item measures self-reported capability rather than actual performance. It includes the functioning of lower extremities (walking or mobility) as well as instrumental activities of daily living, such as running errands. We will use the short form 10b.
  * Physical function, upper extremity: This item measures activities that require use of the upper extremity including shoulder, arm, and hand activities. Examples include writing, using buttons, or opening containers. We will use the short form 7.
  * Pain Interference: This item assesses self-reported consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. We will use the short form 8a.
  Short forms will be used in all sites possible (i.e. where the translation is available).
Patient related outcome / Quality of life 2 | Screening / 6 months follow-up / 12 months follow-up and/or 6 months after bone union (max 18 months)
  EQ-5D-3L assessment (Five items, 3-point categorical scale) The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
  o The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Radiological Outcome | Screening / / Intraoperative / 6 months follow-up / 12 months follow-up and/or 6 months after bone union (max 18 months)
  Pre-operative/intraoperative
  * Deformity parameters (if applicable)
  * Nonunion classification: Hypertrophic, Oligotrophic, Atrophic Follow-up visits
  * Bone healing (based on the treating physician's judgement): Not healed / Partially healed / Mostly healed / Healed
  * Evaluation of the expansion of the bone defect: bone defect size
  * Time to healing: Date when full healing is achieved (to be calculated days from index surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Christoph Pape, MD, Principal Investigator — University Hospital Zurich Department of Trauma Surgery
Locations (21):
- United States (2):
  - Cedar Sinai, Los Angeles, California
  - Sinai Hospital of Baltimore, Baltimore, Maryland
- John Hunter Hospital, Newcastle, Australia
- Hospital Municipal Miguel Couto Serviço de Ortopedia e Traumatologia, Rio de Janeiro, Brazil
- Hospital Base Valdivia, Valdivia, Chile
- Colombia (2):
  - Hospital Universitario de la Samaritana, Bogotá
  - Hospital Pablo Tobon Uribe, Medellín
- Germany (5):
  - University Hospital Frankfurt, Frankfurt
  - Universitätsspital Gießen, Giessen
  - Universitätsklinikum Heidelberg (Unfallchirurgie), Heidelberg
  - Universitätsklinikum Münster (Klinik und Poliklinik für Unfall-, Hand- und Wiederherstellungschirurgie), Münster
  - Krankenhaus Johanneum, Wildeshausen
- Paras HMRI Hospital Patna, Patna, India
- Netherlands (2):
  - Academisch Ziekenhuis Maastricht (Dept. of Surgery), Maastricht
  - Radboud University Medical Center, Nijmegen
- Tygerberg Hospital, Cape Town, South Africa
- Kyungpook National University Hospital (Orthopaedics), Daegu, South Korea
- Universitätsspital Zürich (Klinik für Traumatologie), Zurich, Switzerland
- Central Hospital of Border Guard Service of Ukraine, Kyiv, Ukraine
- Leeds General Infirmary University Hospital (Trauma & Orthopaedic Surgery), Leeds, United Kingdom
- Hospital Universitario de Caracas, Caracas, Venezuela

IPD SHARING:
Plan to Share IPD: Undecided